CLINICAL TRIAL: NCT02435134
Title: Validation of a Test Protocol for Measuring the Hip Internal Rotation Range of Motion Using a Newly Developed Examination Chair
Brief Title: Examination Chair for Hip Internal Rotation Range of Motion Measurement
Acronym: HIRROM
Status: Completed | Type: Observational
Sponsor: Schulthess Klinik (Other)
Responsible Party: Sponsor
Other Study IDs: HIRROM
Record Dates: First submitted 2015-04-27; First posted 2015-05-06 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Limited Hip Mobility

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy participants
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
Hip internal rotation range of motion (HIRROM) assessment is performed to assess the mobility of the hip. The assessment is typically done manually (manual testing), which induces large variability in the results between and within testers. An initial version of an examination chair (EC1) was recently developed with the aim to minimize the variability of testing results for HIRROM assessments. A new version of the examination chair (EC2) has been implemented in order to individualize the testing protocol and will be validated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Participants are pain free in the lower extremity, hip and back
* Participants signed the consent form

Exclusion Criteria:

* Participant requires pain relief medication
* History of hip surgery
* Neuromuscular disorders
* Legal incompetence

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy participants
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-10-07 (Actual); Primary Completion 2017-01-25 (Actual); Study Completion 2017-01-25 (Actual)

PRIMARY OUTCOMES:
Hip internal rotation range of motion angle (degrees) | 7 days
  Participants will be tested for hip internal range of motion using three different methods. The measurements will be repeated 7 days after the initial measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Schulthess Klinik, Zurich, Switzerland